CLINICAL TRIAL: NCT00473902
Title: Creatine Monohydrate and Conjugated Linoleic Acid Improve Strength and Body Composition Following Resistance Exercise in Older Adults
Brief Title: Older Adult Training Study With Creatine and CLA
Acronym: OTR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Older Adult Training Study
Record Dates: First submitted 2007-05-15; First posted 2007-05-16 (Estimated); Last update posted 2007-05-16 (Estimated); Status verified 2007-05

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Creatine; Linoleic Acids, Conjugated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Training
Drug: Creatine Monohydrate, Conjugated Linoleic Acid

SUMMARY:
We examined whether creatine monohydrate (CrM) and conjugated linoleic acid (CLA) could enhance strength gains and improve body composition (i.e., increase fat-free mass (FFM); decrease body fat) following resistance exercise training in older adults (> 65 y). Our study hypothesized that administering CrM and CLA would yield greater strength and body composition benefits than the placebo group over the six months of resistance exercise

DETAILED DESCRIPTION:
Men (N=19) and women (N=20) completed six months of resistance exercise training with Creatine Monohydrate (5g/d) + Conjugated Linoleic Acid (6g/d) or placebo with randomized, double-blind, allocation.Outcomes included; strength and muscular endurance, functional tasks, body composition (DEXA scan), blood tests (lipids, liver function, CK, glucose, systemic inflammation markers (IL-6, C-reactive protein)), urinary markers of compliance (creatine/creatinine), oxidative stress (8-OH-2dG, 8-isoP) and bone resorption (Ν-telopeptides).

ELIGIBILITY:
Inclusion Criteria:

* Healthy,
* Ambulatory,
* Recreationally active,
* Community dwelling

Exclusion Criteria:

* Evidence of coronary heart disease;
* Congestive heart disease;
* Uncontrolled hypertension;
* Chronic obstructive pulmonary disease;
* Diabetes mellitus;
* Renal failure;
* Major orthopedic disability; and
* Smoking

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 39 (Actual)
Dates: Start 2003-08; Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
a. Muscle and bone mass b. Knee extension strength e. Creatine content f. Muscle oxidative capacity g. Aerobic power (oxygen consumption) | six months

SECONDARY OUTCOMES:
a. Functional capacity b. Strength with weight machines | six months

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Tarnopolsky, M.D., Ph.D., Principal Investigator — McMaster University
Locations (1):
- McMaster University Medical Center, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Tarnopolsky M, Zimmer A, Paikin J, Safdar A, Aboud A, Pearce E, Roy B, Doherty T. Creatine monohydrate and conjugated linoleic acid improve strength and body composition following resistance exercise in older adults. PLoS One. 2007 Oct 3;2(10):e991. doi: 10.1371/journal.pone.0000991. PMID 17912368